CLINICAL TRIAL: NCT02263924
Title: Phase III, Single Centre, Double Blind, Randomised, Placebo Controlled, Parallel Group Trial to Evaluate the Efficacy and Safety of Oral Vitamin E (Mixed Tocotrienol) for 6 Months in Patients With Moderate Acute Ischemic Stroke
Brief Title: Stroke and Tocotrienol: Unique Role in Neuroprotection
Acronym: SATURN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seberang Jaya Clinical Research Centre (Other Government)
Collaborators: Clinical Research Centre Hospital Taiping (Unknown); Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-CRC-001-03
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tocotrienols

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either placebo or investigational drug (mixed tocotrienols dietary supplement) for 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Tocotrienol (Experimental): Mixed tocotrienol 200mg twice a day for 6 months
  Interventions: Dietary Supplement: Tocotrienol
- Placebo (for tocotrienol) (Placebo Comparator): Placebo capsules, 1 capsule twice a day for 6 months
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Tocotrienol — Subjects in the intervention arm will take one capsule of 200mg tocotrienol twice daily for 6 months
  Arms: Experimental: Tocotrienol
Dietary Supplement: Placebo capsules — Subjects in the placebo arm will take one capsule of placebo twice daily for 6 months
  Arms: Placebo (for tocotrienol)

SUMMARY:
Phase III, single-centre, double-blind, randomised, placebo-controlled, parallel-group trial to evaluate the efficacy and safety of oral Vitamin E (Mixed Tocotrienol) for 6 months in patients with moderate ischemic stroke.

150 patients will be recruited and randomized to receive either placebo or mixed tocotrienol 200mg twice a day for 6 months. Patients will be followed up and assessed on their functional recovery.

ELIGIBILITY:
Adult patients within 1-10 days ischaemic stroke of moderate severity (NIHSS 6-20)

Inclusion Criteria:

1. Age 35 years old and above.
2. Subject will be included within the time frame of 1-10 days after the first onset of acute cerebral ischaemic stroke with NIHSS between 6 - 20.
3. Subject is neurologically stable after stroke onset, i.e. no fluctuation in clinical conditions.
4. Subject has a modified Rankin Scale from 2-4.
5. Subject has a clinical stroke diagnosis according to WHO stroke diagnosis.
6. Subject is willing to attend at least four sessions of physiotherapy during the study or as deemed needed by the physiotherapist
7. Subjects or his/her legally acceptable representative is willing to provide written informed consent.

Exclusion Criteria:

1. Subject has evidence of intra-cerebral hemorrhage on brain CT scan or MRI
2. Recurrent stroke or previous hospitalisation due to suspected cerebrovascular event.
3. Severe stroke as assessed clinically and/or by appropriate imaging techniques
4. Subject has other significant non-ischemic brain lesion(s) which could affect function or disability.
5. Time of ischemic stroke onset not exactly known
6. Subject has documented underlying medical conditions which may affect assessment or follow-up such as (but not limited to) terminal cancer, liver cirrhosis, severe dementia or psychosis, connective tissue disease, rheumatoid arthritis, severe heart disease, severe liver disease or renal failure (based on recent medical history)
7. Subject has active systemic infection such as (but not limited to) hepatitis and pneumonia
8. Subject has definite indication for full dose or long term anti-coagulation therapy (such as warfarin)
9. Any condition that in the judgment of the investigator would place the patient under undue risk
10. Traumatic brain injury within the previous 30 days.
11. Symptoms which are rapidly improving (as in transient ischemic stroke)
12. The patient is pregnant, breast feeding or female of childbearing potential (unless the subject is willing to practice on double contraception measures for the study duration) until up to 1 month (30 days) after last treatment dose.
13. Patients who have been included in any other clinical trial within the previous three months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Score | 6th Month
  Shift in modified Rankin Score (mRS) at 6 months of treatment (odds ratio)

SECONDARY OUTCOMES:
Modified Rankin Score | 3rd month
  Shift in modified Rankin Score (mRS) at 3 months of treatment (odds ratio)
Modified Barthel Index | 6th months
  • Increment in the score of Modified Barthel Index at the end of 6 months of treatment from baseline (before treatment)
NIHSS | before dosing and at 6th month
  Reduction in NIHSS at the end of 6 months of treatment from baseline
Composite score (MRS, NIHSS, mBI) | 6th month
  Proportion of patients achieving favourable composite score of mRS 0 - 2, NIHSS <6, and mBI at least 95
Modified Rankin Score | 3rd month
  Proportion of patients achieving modified Rankin Score (mRS) of 0 - 2 at 3 months of treatment
Modified Rankin Score | 6th month
  Proportion of patients achieving modified Rankin Score (mRS) of 0 - 2 at 6 months of treatment
MRI - Brain lesion volume | 6th month
  Change in stroke lesion volume
SF-36 | 6th month
  quality of life
CLOX and TMT Parts A & B | 6th month
  Improvement in the score of CLOX and TMT Parts A & B at the end of 24-weeks of treatment from baseline
Adverse event monitoring | 6 months
  Adverse event outcomes in both groups

CONTACTS AND LOCATIONS:
Overall Officials: IRENE LOOI, Principal Investigator — SEBERANG JAYA HOSPITAL CLINICAL RESEARCH CENTRE; KAH HAY YUEN, Study Director — Universiti Sains Malaysia
Locations (1):
- Seberang Jaya Clinical Research Centre, Seberang Jaya, Pulau Pinang, Malaysia